CLINICAL TRIAL: NCT02958696
Title: A Phase 1, Randomised, Open Label, 2-period Crossover, Single Centre, 3-arm, Single Dose Study to Investigate the Relative Bioavailability of HTL0018318 Oral Aqueous Solution Versus Capsule Formation in Healthy Volunteers
Brief Title: Relative Bioavailability of HTL0018318 Oral Aqueous Solution Versus Capsules
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nxera Pharma UK Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HTL0018318-104; 2016-003313-99 (EudraCT Number); 16-024 (Other: HMR Protocol Code)
Record Dates: First submitted 2016-11-01; First posted 2016-11-08 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Bioavailability and Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- HTL0018318 low dose (Active Comparator): low dose aqueous solution and/or equivalent low dose capsule
  Interventions: Drug: HTL0018318
- HTL0018318 mid dose (Active Comparator): mid dose aqueous solution and/or equivalent mid dose capsule
  Interventions: Drug: HTL0018318
- HTL0018318 high dose (Active Comparator): high dose aqueous solution and/or equivalent high dose capsule(s)
  Interventions: Drug: HTL0018318

INTERVENTIONS:
Drug: HTL0018318 — Two single doses of active drug (low, mid or high dose either as aqueous solution or capsule) separated by a washout of at least 12 days.

SUMMARY:
HTL0018318 is a selective muscarinc M1 agonist. This study is a phase I, open label, randomised, crossover, single dose, trial in healthy volunteers to compare the relative bioavailability of HTL0018318 when given by oral aqueous solution and in capsule formulation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female healthy volunteer.
2. Aged 18-55 years.
3. A body mass index (Quetelet index) in the range 18.0-34.
4. Sufficient intelligence to understand the nature of the trial and any hazards of participating in it. Ability to communicate satisfactorily with the investigator and to participate in, and comply with the requirements of, the entire trial.
5. Willingness to comply with the contraception requirements of the trial.
6. Willingness to give written consent to participate after reading the information and consent form, and after having the opportunity to discuss the trial with the investigator or his delegate.
7. Willingness to give written consent to have data entered into The Overvolunteering Prevention System.

Exclusion Criteria:

1. Clinically relevant abnormal history, physical findings, ECG, or laboratory values at the pre-trial screening assessment that could interfere with the objectives of the trial or the safety of the volunteer.
2. QTcF outside range 300-450 msec for males, and 300-470 msec for females at resting ECG at screening and baseline.
3. Family history of unexplained sudden death, or sudden death due to long QT syndrome.
4. Clinically relevant abnormal findings based on 24 h ECG Holter monitoring during screening, including any of the following: > 200 ventricular ectopic heart beats, ventricular tachycardia, defined as >= 3 successive ventricular ectopic beats at a rate of >120 bpm, second degree heart block, sustained cardiac arrhythmias, including atrial fibrillation, complete heart block and supraventricular tachycardia (SVT), any symptomatic arrhythmia except isolated extra systoles.
5. Aspartate transaminase (AST), alanine transaminase (ALT), gamma glutamyl transferase (GGT) or total bilirubin >1.5 x ULN at screening, or other laboratory blood chemistry test results outside the normal reference range unless deemed not clinically significant by the investigator.
6. Clinically significant renal insufficiency as indicated by a glomerular filtration rate lower than the age-related L at screening. In the event of a glomerular filtration rate >80, eligibility may be confirmed by a second measurement.
7. Blood pressure and heart rate in supine position at the screening examination outside the ranges 90-140 mm Hg systolic, 50-90 mm Hg diastolic; heart rate 45-100 beats/min. Subject with borderline values can be included if the values are deemed not clinically significant by the investigator.
8. Presence of acute or chronic illness or history of chronic illness sufficient to invalidate the volunteer's participation in the trial or make it unnecessarily hazardous.
9. Impaired gastrointestinal, endocrine, thyroid, hepatic, cardiovascular, respiratory, haematological, renal or neurological function, diabetes mellitus, coronary heart disease, or history of any psychotic mental illness deemed clinically significant by the investigator.
10. History of a chronic respiratory condition, such as asthma, recurrent chest infections of chronic obstructive pulmonary disease.
11. History of epilepsy or seizures.
12. History of a severe allergy. Non-active hayfever is acceptable.
13. Surgery (e.g. stomach bypass) or medical condition that might affect absorption, metabolism or elimination of medicines.
14. Presence or history of severe adverse reaction to any drug.
15. Woman who is pregnant or lactating, or pre-menopausal woman who is sexually active and not using a reliable method of contraception.
16. Use of a prescription or over-the-counter medicine, or any herbal remedy or nutritional supplement, during the 21 days before the first dose of trial medication until the end of the study, with the exception of acetaminophen (paracetamol), hormonal contraceptives or hormone replacement therapy (HRT).
17. Presence or history of drug or alcohol abuse in the last 5 years, or intake of more than 21 units of alcohol weekly (for men) or 14 units of alcohol weekly (for women), or use of cigarettes or nicotine-containing products during the 3 months before the first dose until the end of the study.
18. Evidence of drug abuse on urine testing.
19. Positive test for hepatitis B, hepatitis C or HIV.
20. Positive test for alcohol or smoking before dosing.
21. Participation in another clinical trial of a new chemical entity or a prescription medicine within the previous 3 months.
22. Loss of more than 500 mL blood during the 3 months before the trial, eg as a blood donor.
23. Possibility that the volunteer will not cooperate with the requirements of the protocol.
24. Objection by General Practitioner (GP) to volunteer entering trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2016-10; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of HTL0018318 | Predose to 168h post dose
  Comparison of bioavailability in plasma
Area under the curve (AUC) of HTL0018318 | Predose to 168h post dose
  Comparison of bioavailability in plasma

SECONDARY OUTCOMES:
Time to maximum concentration (tmax) | Predose to 168h post dose
  Pharmacokinetics in plasma
Half-life (t1/2) | Predose to 168h post dose
  Pharmacokinetics in plasma
Apparent volume of distribution (Vz/F) | Predose to 168h post dose
  Pharmacokinetics in plasma
Apparent clearance (CLp/F) | Predose to 168h post dose
  Pharmacokinetics in plasma
Amount excreted in urine (Ae) | Predose to 168h post dose
  Pharmacokinetics in urine
Fraction excreted in urine (fe/F) | Predose to 168h post dose
  Pharmacokinetics in urine
Clearance in urine (CLr) | Predose to 168h post dose
  Pharmacokinetics in urine
Treatment-emergent adverse events | Predose up to 28 days post dose
  Adverse events
Vital signs | Predose up to 28 days post dose
  Heart rate and blood pressure
Physical examinations | Predose up to 28 days post dose
  Physical examinations
Laboratory safety assessments | Predose up to 28 days post dose
  Hematology
ECG | Predose up to 28 days post dose
  ECG

CONTACTS AND LOCATIONS:
Overall Officials: Adeep Puri, MPhil MBBS, Principal Investigator — Hammersmith Medicines Research
Locations (1):
- Hammersmith Medicines Research, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No